CLINICAL TRIAL: NCT02119013
Title: EFFECT OF SOMATOSTTIN ON EARLY DIASTOLIC LEFT VENTRICULAR FUNCTION IN AUTOSOMAL DOMINANT POLYCYSTIC KIDNEY DISEASE: A MATCHED-COHORT, SPECKLE-TRACKING ECHOCARDIOGRAPHIC STUDY
Brief Title: Effects of Somatostatin on ADPKD Heart
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADPKD-heart
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; Glomerular Filtration Rate > 40 ml/Min
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCTEOTRIDE (Experimental): Octeotride, 20 mg monthly intramuscular injection for 3 years
  Interventions: Drug: Octeotride
- PLACEBO (Placebo Comparator): Placebo (salin soluction), intramuscular injection monthly for 3 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octeotride
  Arms: OCTEOTRIDE
Drug: Placebo
  Arms: PLACEBO

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is associated with early onset hypertension and left ventricular (LV) hypertrophy. Since LV hypertrophy is associated with LV diastolic function impairment, we aimed to assess the changes over time of LV diastolic function in ADPKD patients and whether they were affected by the treatment with the somatostatin analogue, octreotide.

35 ADPKD patients (14 males) aged 34±8 years (mean glomerular filtration rate 82±26 mL/min/1.73m2) were randomly assigned to 36 month treatment with placebo (n=18) or octreotide (n=17). Clinical and echocardiography parameters were evaluated at baseline and study end. LV mass (M) and ejection fraction (EF) were calculated according to Devereux formula and biplane Simpson's algorithm, respectively. LV filling was assessed by mitral and pulmonary vein flow velocity curves and mitral annulus early diastolic velocity peak (Ea) by tissue Doppler imaging.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autosomal dominant polycystic kidney disease
* glomerular filtration rate grater than 40 ml/min

Exclusion Criteria:

* diabetes mellitus
* proteinuria greater than 1 g/24 hours
* significant glomerular disease
* urinary tract lithiasis and infections
* symptomatic gallstones
* biliary sludge
* cancer
* pregnant women
* lactanting women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
EFFECT ON LEFT VENTRICULAR DYASTOLIC FUNCTION | 3 years
  To assess the changes over time of left ventricular dyastolic function in ADPKD patients and whether they were affected by the treatment with the somatostatin analogue, octreotide

CONTACTS AND LOCATIONS:
Overall Officials: eleonora riccio, md, Principal Investigator — Federico II University